CLINICAL TRIAL: NCT00613886
Title: Factors Predicting Response to Shunting in Normal Pressure Hydrocephalus
Acronym: NPH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was withdrawn as number of subjects enrolled did not meet expectation
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS 2005-4609; J&J Proposal #38973 (Other: J&J Proposal #38973); Award #032906 (Other: Award #032906)
Record Dates: First submitted 2008-01-03; First posted 2008-02-13 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: NPH; Normal Pressure Hydrocephalus
MeSH Terms: conditions — Hydrocephalus, Normal Pressure | interventions — Physical Therapy Modalities; Occupational Therapy; Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Comparison for patients of lumbar drain and shunt surgery (Experimental): Subjective comparisons made for patients - before and after external lumbar drain, before and after shunt surgery.
  Device: Programmable Shunt Insertion (Codman Medtronic)
  Behavioral: Assessments in physical therapy, occupational therapy, and speech therapy
  Follow-up testing to be administered by trained physician assistant in the outpatient setting on an approximately monthly basis: 10m walk, timed up-and-go, mini-mental status exam, 9-hole grooved pegboard, motor visual perception test (MVPT), modified rankin score (MRS)
  Interventions: Device: Programmable Shunt Insertion (Codman, Medtronic); Behavioral: Assessments in physical therapy, occupational therapy, and speech therapy

INTERVENTIONS:
Device: Programmable Shunt Insertion (Codman, Medtronic) — Medical Device - Shunt insertion surgery of adjustable valve and laparoscopic assistance for placement of peritoneal catheter. Patient will be brought to operating room suite where general anesthesia is induced. Patient will be placed with a small roll on shoulder, supine, on the operating room table. Patient's head will be turned with the parietal area uppermost in the field. Patient will be prepared and draped in the usual sterile fashion. Site prep includes parietooccipital area, side of neck, chest, and entire abdomen. Ventricular catheter placed and then attached to shunt valve. Catheter is then fitted over grooved blue burr hole guide. Excess catheter pulled down to pull valve into pocket on the skull. Sterile dressings applied.
  Other Names: Codman Shunt; Medtronic Strata Valve
Behavioral: Assessments in physical therapy, occupational therapy, and speech therapy — Follow-up testing to be administered by trained Physician Assistant in the outpatient setting on an approximately monthly basis: 10m walk, timed up-and-go, Mini-Mental Status Exam, 9-hole Grooved Pegboard, Motor Visual Perception Test (MVPT), Modified Rankin Score (MRS)

SUMMARY:
The research project is designed to determine which combination of tests will enable physicians to predict whether a patient with symptoms of normal pressure hydrocephalus (NPH) will improve with a shunt.

DETAILED DESCRIPTION:
Normal pressure hydrocephalus (NPH) is a potentially reversible progressive neurological condition disproportionately affecting the elderly population. Given current controversies regarding its exact definition, accurate incidence and prevalence figures are elusive. NPH was first described forty years ago as a triad of symptoms consisting of gait difficulties, urinary incontinence, and memory problems in patients with enlarged ventricles in the absence of increased intracranial pressure (ICP). The cause of primary, or idiopathic NPH (INPH) remains elusive, while secondary NPH results from intracranial insults such as head trauma, meningitis, or intracranial hemorrhage. NPH can be successfully treated with cerebrospinal fluid (CSF) shunting. However, the accurate diagnosis and treatment of patients with NPH remains problematic, despite significant advances in brain imaging and ICP physiology.

Objectives - The primary aims of this study are:

1. to confirm the ability of external lumbar drainage to increase the success rate of selectively shunting patients with NPH compared to historical controls
2. to refine the diagnosis of NPH by determining whether the factors that change before and after lumbar drainage will predict failure to improve after shunting. A related aim is to assess the complications attributable to lumbar drainage.
3. to perform a preliminary evaluation of programmable shunt valves for NPH compared to historical controls using fixed-pressure valves. A related aim is to determine whether post-op objective analysis of gait, cognitive function and urinary symptoms will help refine the programmable shunt setting on an individual basis.

Secondary study aims include:

Investigating the pathophysiology of NPH by: 1) correlating cortical vein compliance measured by MRI flow quantification studies with CSF pressure waveform analysis; 2)assessing funduscopic changes before and during ELD; 3) performing and cross correlating CSF chemical analysis on screening positive and negative patients as well as screening-positive patients who are shunt responsive versus unresponsive.

ELIGIBILITY:
Inclusion Criteria:

* Walking difficulties in both legs which has developed gradually, not explained by other conditions, either in combination with mental impairment and urinary incontinence
* Brain CT or MRI findings of enlarged ventricles compared to established standards (minimum Evans ratio of 0.30 as measured by reviewing films)
* Mental impairment must be mild to moderate, emerging with or after the walking difficulties
* Age > or = 18 years old
* MMSE (Mini-mental status exam): < or = 10
* Urinary incontinence

Exclusion Criteria:

* No or only minimal walking difficulties combined with severe dementia
* Severe medical problems with limited life expectancy (less than six months)
* Contraindications to surgery
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Pare, MD, FRCSC, Principal Investigator — UC Irvine
Locations (1):
- University of California, Irvine - Medical Center, Orange, California, United States

REFERENCES:
- See also: UC, Irvine Medical Center - Dept of Neurosurgery's NPH webpage — http://neurosurgery.uci.edu/nph_article.shtml

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With External Lumbar Drain and Shunt Surg: All NPH patients shunted under this protocol have had a programmable valve inserted, either the Medtronic Strata valve, or the Codman-Hamim programmable valve. The valve pressure is set at the highest opening pressure at the time of implantation
Period: Overall Study
Arm/Group | Patients With External Lumbar Drain and Shunt Surg
Started | 24
Completed | 0
Not Completed | 24

BASELINE CHARACTERISTICS:
Population: Subjects enrolled
Groups:
- Subjective Comparisons Made for Patients - Before and After ex: Programmable Shunt Insertion (Codman, Medtronic): Medical Device - Shunt insertion surgery of adjustable valve and laparoscopic assistance for placement of peritoneal catheter. Patient will be brought to operating room suite where general anesthesia is induced. Patient will be placed with a small roll on shoulder, supine, on the operating room table. Patient's head will be turned with the parietal area uppermost in the field. Patient will be prepared and draped in the usual sterile fashion. Site prep includes parietooccipital area, side of neck, chest, and entire abdomen. Ventricular catheter placed and then attached to shunt valve. Catheter is then fitted over grooved blue burr hole guide. Excess catheter pulled down to pull valve into pocket on the skull. Sterile dressings applied.
  Assessments in physical therapy, occupational therapy, and speech therapy:
Arm/Group | Subjective Comparisons Made for Patients - Before and After ex
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Evans Ratio
Description: A brain CT scan is obtained after the first week to ten days and the shunt is adjusted according to the patients signs and symptoms. Prior to any downward adjustment of the shunt valve (which allows more CSF drainage), a brain CT is obtained to look for subdural hematoma or effusion. If any type of subdural collection is found, the valve pressure is increased (to reduce CSF flow) until the collection resolves.
Time Frame: initial and follow-up visits
Population: Insufficient number of participants were recruited to conduct qualitative analysis. The PI ended recruitment and left the university therefore no study data was produced.
Groups:
- Comparison for Patients of Lumbar Drain and Shunt Surgery: Subjective comparisons made for patients - before and after external lumbar drain, before and after shunt surgery.
  Device: Programmable Shunt Insertion Behavioral: Assessments in physical therapy, occupational therapy, and speech therapy Follow-up testing to be administered by trained physician assistant in the outpatient setting on an approximately monthly basis: 10m walk, timed up-and-go, mini-mental status exam, 9-hole grooved pegboard, motor visual perception test (MVPT), modified rankin score (MRS) Programmable Shunt Insertion (Codman, Medtronic): Medical Device - Shunt insertion surgery of adjustable valve and laparoscopic assistance for placement of peritoneal catheter.
Arm/Group | Comparison for Patients of Lumbar Drain and Shunt Surgery
Number analyzed (Participants) | 0

2. Secondary Outcome: Physical Therapy, Occupational Therapy, and Speech Therapy
Description: The evaluations for physical therapy, occupational therapy and speech therapy are performed along with external lumbar drainage (ELD) to assess NPH subjects.
Time Frame: 30 min per clinic visit
Population: Insufficient number of subjects recruited for significant analysis. The PI ended recruitment and left the university therefore no study data was produced.
Groups:
- Comparison for Patients of Lumbar Drain and Shunt Surgery: Subjective comparisons made for patients - before and after external lumbar drain, before and after shunt surgery.
Arm/Group | Comparison for Patients of Lumbar Drain and Shunt Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Comparison for Patients of Lumbar Drain and Shunt Surgery: Subjective comparisons made for patients - before and after external lumbar drain, before and after shunt surgery.
  Device: Programmable Shunt Insertion (Codman Medtronic) Behavioral: Assessments in physical therapy, occupational therapy, and speech therapy Follow-up testing to be administered by trained physician assistant in the outpatient setting on an approximately monthly basis: 10m walk, timed up-and-go, mini-mental status exam, 9-hole grooved pegboard, motor visual perception test (MVPT), modified rankin score (MRS) Programmable Shunt Insertion(Codman, Medtronic): Medical Device - Shunt insertion surgery of adjustable valve and laparoscopic assistance for placement of peritoneal catheter.
Arm/Group | Comparison for Patients of Lumbar Drain and Shunt Surgery
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No